CLINICAL TRIAL: NCT00745225
Title: Targeting Peroxisome Proliferator-Activated Receptor-Gamma in Peritoneal Dialysis Patients - Will it Reduce Inflammation, Atherosclerosis, Calcification and Improve Survival of Peritoneal Dialysis Patients? (PROOF Trial)
Brief Title: Peroxisome Proliferator-Activated Receptor-Gamma Activation in Peritoneal Dialysis Patients
Acronym: PPAR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Principal Investigator, Dr. Angela Yee-Moon Wang, Dr., The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A111-101
Record Dates: First submitted 2008-09-01; First posted 2008-09-03 (Estimated); Last update posted 2021-10-08 (Actual); Status verified 2021-10

CONDITIONS: End-stage Renal Disease
Keywords: peritoneal dialysis, cardiovascular, PPAR-gamma
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Pioglitazone

STUDY DESIGN:
Intervention Model Description: Double-blind randomized placebo-controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind randomized placebo-controlled trial, all parties are masked
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active intervention arm (Experimental): Peroxisome proliferator activator receptor gamma treatment, Pioglitazone
  Interventions: Drug: Pioglitazone
- placebo pill (Placebo Comparator): placebo comparator
  Interventions: Drug: placebo comparator

INTERVENTIONS:
Drug: Pioglitazone — pioglitazone 15mg daily for 12 weeks, then 30mg daily for 84 weeks
  Other Names: Actos
  Arms: Active intervention arm
Drug: placebo comparator — 1 capsule daily, 96 weeks.
  Other Names: Placebo
  Arms: placebo pill

SUMMARY:
To study whether peroxisome proliferator-activated receptor-gamma activation in peritoneal dialysis patients will reduce inflammation, atherosclerosis, calcification and improve survival of peritoneal dialysis patients

DETAILED DESCRIPTION:
Peritoneal dialysis patients are at increased risk of cardiovascular morbidity and mortality and are related to the presence of accelerated atherosclerosis. Other than the traditional cardiovascular risk factors, there is increasing evidence that inflammation is associated with the development of atherosclerosis and cardiovascular events in both the general and dialysis population. C-reactive protein is predictive of higher all-cause mortality and cardiovascular mortality, independent of other cardiovascular risk factors and atherosclerotic vascular disease. As a considerable proportion of peritoneal dialysis patients showed elevated C-reactive protein, it raises an important question as to whether lowering C-reactive protein will have any cardiovascular and survival benefit in these patients. On the other hand, insulin resistance with associated hyperinsulinemia is frequently observed in chronic renal failure and dialysis patients. Although the exact mechanism of insulin resistance needs further evaluation, studies indicated that insulin resistance is an important cardiovascular risk factor and outcome predictor in the general and dialysis population. Moreover, recent evidence indicates an association between chronic inflammation and insulin resistance although the exact interrelationship remains unclear. The peroxisome proliferator-activated receptor-gamma (PPAR-g) is a member of the nuclear receptor family of ligand-dependent transcription factors. PPAR-g is highly expressed in adipose tissue and clinical study has confirmed efficacy of the specific ligands for PPAR-gamma, namely thiazolidinediones (TZD), in improving insulin sensitivity. Recent experimental and clinical studies demonstrated that TZD has anti-inflammatory and anti-atherosclerotic properties other than insulin sensitizing effect in type 2 diabetics. We hypothesize that modulation of the PPAR-g activity may be a novel therapeutic strategy for reducing inflammation and improving insulin sensitivity and may retard the progression of atherosclerosis and possibly reduce mortality of our peritoneal dialysis patients.

ELIGIBILITY:
Inclusion Criteria:

* Both prevalent patients or patients newly started on continuous peritoneal dialysis, with or without diabetes mellitus will be considered eligible for study entry.
* For patients newly started on chronic peritoneal dialysis, they will be suitable for recruitment into the study after one month on peritoneal dialysis.
* Patients who provide informed consent for the study

Exclusion Criteria:

* Patients with underlying active malignancy
* Patients with chronic liver disease or liver cirrhosis
* Patients with active infections
* Patients with other chronic active inflammatory disease such as systemic lupus erythematosus, rheumatoid arthritis
* Patients who refuse study participation
* Patients with underlying congenital heart disease or rheumatic heart disease
* Patients with poor general condition
* Patients with plans for living related kidney transplant within 2 years
* Female patients with pregnancy
* Patients with history of recurrent hypoglycemia
* Patients with Class III and IV congestive heart failure
* Patients already receiving glitazones treatment at the screening visit

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2006-02 (Actual); Primary Completion 2014-10 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Change in carotid intima-media thickness | over 48 weeks
  Change in carotid intima-media thickness
change in flow mediated dilatation (marker of endothelial function) | over 48 weeks
  change in flow mediated dilatation (marker of endothelial function)

SECONDARY OUTCOMES:
change in aortic pulse wave velocity | over 96 weeks
  change in aortic pulse wave velocity
change in augmentation index-heart rate adjusted | over 96 weeks
  change in augmentation index-heart rate adjusted
change in nitroglycerin-mediated dilatation | over 48 weeks
  change in nitroglycerin-mediated dilatation
change in coronary artery calcium score | over 96 weeks
  change in coronary artery calcium score
change in heart valves calcium score | over 96 weeks
  change in heart valves calcium score
change in carotid artery calcium score | over 96 weeks
  change in carotid artery calcium score
change in abdominal visceral fat | over 96 weeks
  change in abdominal visceral fat
change in subcutaneous fat | over 96 weeks
  change in subcutaneous fat
change in blood pressure | over 96 weeks
  change in blood pressure
change in C-reactive protein | over 96 weeks
  change in C-reactive protein
change in residual kidney function | over 96 weeks
  change in residual kidney function
change in HOMA index (among those not on insulin) | over 96 weeks
  Change in insulin resistance index
change in D/P creatinine ratio | over 96 weeks
  Change in peritoneal solute transport parameter
change in peritoneal ultrafiltration with 2.5% during PET | over 96 weeks
  Change in peritoneal ultrafiltration volume
change in handgrip strength | over 96 weeks
  change in handgrip strength
Change in cardiac biomarkers | over 96 weeks
  change in cardiac biomarkers
change in insulin dose (among those on insulin) | over 96 weeks
  change in insulin dose
change in endothelial progenitor cells | over 96 weeks
  change in endothelial progenitor cells
change in central systolic blood pressure | over 96 weeks
  change in central systolic blood pressure
Change in central diastolic blood pressure | over 96 weeks
  change in central diastolic blood pressure
change in glycemic control (fasting glucose, and glycosylated hemoglobin) | over 96 weeks
  change in glycemic control

OTHER OUTCOMES:
overall survival | over 96 weeks
  Hard outcome
major adverse cardiovascular event-free survival | over 96 weeks
  hard outcome
Fluid overload/heart failure event-free survival | over 96 weeks
  hard outcome
myocardial infarction event-free survival | over 96 weeks
  hard outcome
3 point major adverse cardiovascular event-free survival | over 96 weeks
  Hard outcome
4 point major adverse cardiovascular event-free survival | over 96 weeks
  Hard outcome

CONTACTS AND LOCATIONS:
Overall Officials: Angela YM Wang, MD, PhD, FRCP, Principal Investigator — University of Hong Kong, Queen Mary Hospital
Locations (1):
- Queen Mary Hospital, Tung Wah Hospital, Hong Kong, Hong Kong